CLINICAL TRIAL: NCT06341244
Title: Air Stacking Technique Efficacy on Expiratory Peak of Expiratory Flow and Cough Peak Flow in Patients Undergoing Non-cardiac Thoracic Surgery
Brief Title: Air Stacking Technique Efficacy on Peak of Expiratory Flow and Cough Peak Flow in Non-cardiac Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luciana Chiavegato, PhD, Universidade Cidade de Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIFESP
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Care
Keywords: Physiotherapy; Cough; Peak Expiratory Flow
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air staking technique group (Experimental): The air staking group
  Interventions: Device: Air Stacking Technique

INTERVENTIONS:
Device: Air Stacking Technique — To perform the air stacking technique, an air manual breathing unit (AMBU) was used, attached to a unidirectional valve and nasal/oral mask. For each AMBU manual compression (three in the total), the patient was instructed to breathe in deeply and hold the air inside the lungs.

SUMMARY:
After thoracic surgical intervention, patients often feel intense pain with respiratory movements reduction making coughing less effective. The air stacking improves peak of expiratory flow (PEF) and cough peak flow (CPF) in neuro myopathies, thus raising the hypothesis that may also be effective in patients undergoing thoracic surgeries. Objectives: To evaluate the effectiveness, safety and feasibility of air stacking on postoperative PEF and CPF in patients undergoing thoracic surgeries. Methods: Patients undergoing thoracic surgery underwent air stacking on 3th PO. Dyspnea, pain, SpO2, maximum inspirational pressure (MIP), maximum expiratory pressure (MEP), PEF and CPF were evaluated in pre and postoperatory.

DETAILED DESCRIPTION:
Surgical intervention is a treatment option for many diseases of the thorax . After thoracotomy, ventilatory patterns change, lung volumes and pulmonary capacities decrease due to the reflex inhibition of the diaphragm muscle, and the sigh mechanism becomes impaired, even if the procedure does not include pulmonary resection . These changes often lead to postoperative pulmonary complications, which may increase length of stay in the hospital. The role of physical therapy in minimizing these risks is critical, and several techniques are available to improve both lung volume and capacity and to make coughing more effective. The air stacking technique allows enough air to be accumulated in the lungs to generate an acceptable cough peak flow (CPF). Several studies have shown that the use of this technique in patients with neuromuscular disease positively impacts the biomechanical components of peak expiratory flow (PEF) and CPF. This study aimed to evaluate the effectiveness, safety and feasibility of the air stacking technique application and its effect on PEF and CPF during the postoperative period in patients undergoing elective noncardiac intrathoracic surgery We conducted an interventional experimental study involving hospitalized patients for thoracic surgery in a teaching hospital. The study was approved by the Ethics Committee in Human Research (42693015.0.000.5505), and the patients freely signed an informed consent form prior to participation. Maximal inspiratory and expiratory pressure (MIP and MEP) were measured with a previously calibrated aneroid manometer (GER-AR®), ranging from 5 to ± 300 cmH2O. A mouthpiece was attached to the manovacuometer, and the nasal clip was used during the maneuvers following previous recommendations. (12) For maximal inspiratory and expiratory pressures assessment, maximum effort was requested from the residual volume and total lung capacity, respectively. Results were compared to predicted values according to the equation proposed by Neder et al. PEF and CPF were measured with a peak flow meter ranging from 100 to 900 L/min following the literature recommendations. The patient remained seated at 90º with a nasal clip and was asked to force maximum expiration as fast as he could through the mouthpiece after maximum inspiration to measure PEF. To measure cough peak flow, the patient repeated the inspiratory maneuver and was asked to cough as hard as he could. At least three measurements of both variables were performed, provided that the last measurement was not higher than others. The highest obtained value was considered as the result. To perform the air stacking technique, an air manual breathing unit (AMBU) was used, attached to a unidirectional valve and nasal/oral mask. The technique was performed with the patient in a sitting position, head resting on a smooth surface to avoid neck hyperextension. The mask was fit to the patient's face, and the AMBU one-way valve was kept closed. For each AMBU manual compression (three in the total), the patient was instructed to breathe in deeply and hold the air inside the lungs. Immediately after the first manual compression, the second and third were performed while the patient is deep breathing in together, without exhaling the air. PEF was measured immediately after the technique. The patient rested for 5 minutes, and the air staking technique was repeated. The same procedure was performed to measure CPF followed by a clinical evaluation including vital signs, visual lung expansion and auscultation, dyspnea, and pain evaluation. Sample size calculation was based on previous study performed by Brito et al. A minimum difference of 4% and a maximum difference of 47% were found between PEF and CPF means before and after air stacking technique. Considering a power of 90% and an alpha error of 5%, a power analysis revealed that a minimum number of 17 patients should be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older eligible for elective noncardiac intrathoracic surgery;
* Any gender;
* Clinically stable
* Able to perform study procedures.

Exclusion Criteria:

* Patients remained on mechanical ventilation for more than 72 hours at the PO;
* Rib fracture
* Rehospitalization in the ICU or readmission to the intensive care unit (ICU);
* Lowed level of consciousness, nausea and vomiting;
* Hemodynamic instability;
* New surgical intervention before the 3rd.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Peak of expiratory flow (PEF) | pre operative and 3th postoperative day ( pre and pos air stacking application)
  PEF was measured with a peak flow meter ranging from 100 to 900 L/min (Philips Respironics®) following the literature recommendations. The patient remained seated at 90º with a nasal clip and was asked to force maximum expiration as fast as he could through the mouthpiece after maximum inspiration to measure PEF
Cough peak flow (CPF) | pre operative and 3th postoperative day ( pre and pos air stacking application)
  CPF were measured with a peak flow meter ranging from 100 to 900 L/min (Philips Respironics®) following the literature recommendations. The patient remained seated at 90º with a nasal clip and was asked to force maximum expiration as fast as he could through the mouthpiece after maximum inspiration to measure PEF. To measure cough peak flow, the patient repeated the inspiratory maneuver and was asked to cough as hard as he could. At least three measurements of both variables were performed

SECONDARY OUTCOMES:
Maximum Inspiratory Pressure ( MIP) | pre operative and 3th postoperative day ( pre and pos air stacking application)
  MIP and MEP) were measured with a previously calibrated aneroid manovacuometer (GER-AR®), ranging from 5 to ± 300 cmH2O. A mouthpiece was attached to the manovacuometer, and the nasal clip was used during the maneuvers following previous recommendations
Maximun Expiratory Pressure (MEP) | pre operative and 3th postoperative day ( pre and pos air stacking application)
  MIP and MEP) were measured with a previously calibrated aneroid manovacuometer (GER-AR®), ranging from 5 to ± 300 cmH2O. A mouthpiece was attached to the manovacuometer, and the nasal clip was used during the maneuvers following previous recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Luciana D Chiavegato, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Luciana Chiavegato, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The pre operative evaluation records are available in a box kept in the private hospital specific room.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data been available since the beginning and will be until the study publication
Access Criteria: All researchers involved will have access to the hospital private room and data